CLINICAL TRIAL: NCT05404022
Title: Cancer Behavioural Nutrition and Exercise Feasibility Trial - Phase II Randomised Controlled Trial Among Older Adults With Lung Cancer
Brief Title: Feasibility Trial of a Personalised Nutrition and Activity Programme for People With Lung Cancer Over 65 Years
Acronym: CanBenefitII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RS166
Record Dates: First submitted 2022-05-12; First posted 2022-06-03 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2022-06

CONDITIONS: Lung Neoplasm Malignant; Mesothelioma; Lung
Keywords: Physical Activity; Nutrition; Feasibility RCT; Lung cancer; Older adults
MeSH Terms: conditions — Lung Neoplasms; Mesothelioma; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): 12 weeks home based tailored nutrition and physical activity (PA) programme Participants will have an appointment (face-to-face if possible) with the study physiotherapist and dietitian for delivery of the PA (including breathlessness management) and nutrition intervention components. Participants will receive study equipment at these appointments (or by post) including paper-based tracking diary, resistance bands for strength exercises, a Fitbit activity monitor to track steps and aerobic activity during the study period, nutritional supplements (if prescribed), and printed study materials (if preferred over pdf emails; e.g. cooking tips, recipes). A video/telephone follow-up call (10-15 minutes) will be conducted by the research team with the participant at weeks 2,3,4,5 and 6 and then at weeks 8,10 and 12 to review and adjust their programme (with input from the physiotherapist and dietitian if required).
  Interventions: Other: Tailored nutrition and physical activity programme
- Usual care arm (No Intervention): The usual cancer care will include usual patient management and care prior, during and after cancer treatment - medication, symptom control, cancer advice and support from routine medical and nursing input with access to Allied Health Professionals (AHPs) such as physiotherapists and dietitians as clinically indicated. As part of this, it is common for older adults with cancer to be prescribed high protein supplementation. Control participants will receive a general information leaflet regarding activity and nutrition.

INTERVENTIONS:
Other: Tailored nutrition and physical activity programme — Physical activity prescriptions will follow recent guidance for people with cancer and the FITT principles: Frequency (weekly sessions), Intensity (how hard), Time (session duration), and Type. Programme content, duration, and intensity will be tailored for comorbidities and other limitations.
  Nutrition prescription may include any or all of the following:
  1. Information on side-effects that may affect eating and their mitigation
  2. Feedback on physical measures (weight loss) in relation to nutrition and treatment outcomes
  3. Feedback on assessment of food intake and how to improve
  4. a Macmillan booklet: advice on eating and maintaining weight throughout cancer treatments.
  5. a recipe book "Making the most of every bite"
  6. tailored oral nutritional support, including use of high calorie/protein nutrition supplementation, or other macro and micronutrient supplementation as required
  Arms: Intervention arm

SUMMARY:
People with cancer affecting the lungs tend to be older and frailer compared to people with other cancers. As a result, they may have poorer quality of life and are less able to tolerate treatments for their cancer, such as chemotherapy. Research to date show that nutrition and physical activity support helps people with cancer, but not many older people are included in these studies.

The investigators want to develop and test a nutrition and activity programme for older people with lung cancer that can be tailored to each patient to help them have the best possible quality of life from the moment they start a new line of cancer treatment.

The research team has conducted the development work to find which nutrition and activity programmes are best for this patient group and how best to deliver the programme by looking at prior studies and talking to patients and carers as well as health care providers.

The next step is to test the developed programme in a small pilot study, to i) see if it is possible and acceptable (to patients, families, and staff) to deliver and ii) see if it helps patients have and cope with anti-cancer treatments and improve patient quality of life.

DETAILED DESCRIPTION:
BACKGROUND

Lung cancer is the third most commonly diagnosed cancer in the UK and most common in Yorkshire. It is also the most common cause of cancer death in UK. People with lung cancer are often older with co-morbidities and frailty resulting in a poor prognosis - especially if they are unfit for treatment. Approximately half of new cancer cases in UK are people aged 65 and over. Frailty, with sarcopenia (age-related decline in skeletal muscle), cachexia (disease-related body wasting) and nutritional deficiencies, may limit chemotherapy options, reduce treatment effectiveness, result in dose reductions and poor treatment completion rates.

Physical activity (PA) interventions benefit people living with or beyond cancer by improving physical function and quality of life (QoL) during and after cancer treatment. Reduced physical function is associated with higher mortality in older adults with cancer.PA improves treatment completion, treatment recovery, survival rates and reduces healthcare use. Emerging work indicates that activity improves immune function in older adults with cancer; important as better immune function has been linked to improved treatment outcomes. A recent meta-analysis shows reduced risk of cancer-specific and all-cause mortality for those more active among people with lung cancer.

Weight loss and poor nutrition may prevent patients from completing cancer treatments and increase the risk and severity of treatment toxicity. In those receiving chemotherapy, better nutritional status is associated with improved survival and, in lung cancer patients undergoing chemotherapy, better QoL. Cancer treatments can cause many side-effects that impact eating, including; fatigue, nausea, vomiting, dry mouth/oral candidiasis, disordered taste, ill-fitting dentures, diarrhoea, constipation, oesophagitis, early satiety and poor appetite; all difficult for patients to self-manage. Nutritional interventions, including dietary counselling and nutrition advice, improve patient wellbeing and rate of treatment completion. Despite the urgent need for improvements in survival outcomes for older people with lung cancer, a significant evidence gap remains regarding nutrition.

This team's systematic review highlighted the lack of PA and nutrition programme research for older adults living with and beyond cancer. Studies including older adults often focus on prostate cancer, generally a group with a better prognosis. Therefore, many older adults with other cancers, such as lung cancer (only one study in our review), are not represented. Qualitative interviews with patients, carers, and clinicians in Hull (with experience of lung cancer) confirmed poor access to, but support for and interest in, wellbeing interventions but only if tailored to their needs - including management of activity-related breathlessness.

A tailored wellbeing intervention, designed to improve or maintain physical function via lifestyle behaviours, may decrease older adults with lung cancer needing dose reductions. Dose intensity is significantly associated with mortality among people receiving treatment for lung cancer. By maintaining physical function/nutrition, people can tolerate more treatment with subsequent better overall survival. This could be very significant among people diagnosed with lung cancer, a cancer with generally poor prognosis.

Therefore, the aim of this study is to investigate the feasibility and acceptability of conducting a future definitive trial of a tailored wellbeing (nutrition and activity) programme for older adults with lung cancers who are starting a new line of systemic anticancer therapy.

AIMS AND OBJECTIVES

Primary aim/objective

To determine the feasibility and acceptability of a tailored wellbeing (nutrition and activity) programme for older adults with lung cancer beginning a new line of systemic anti-cancer therapy in terms of recruitment, intervention delivery, appropriateness of candidate primary outcomes, estimated sample size for a future phase III trial.

Secondary aims/objectives

To assess data quality

1. QoL* and QoL adjusted days alive out of hospital*
2. treatment dose intensity*
3. episodes of infection
4. fatigue
5. functional status

To assess participant/clinician acceptability and experience

*candidate primary outcomes for subsequent trial

ELIGIBILITY:
Inclusion Criteria:

1. age ≥65 years,
2. diagnosed with stage III or IV lung cancer or mesothelioma,
3. starting a new line of systemic anti-cancer treatment,
4. willing and able to complete study measures and be randomised
5. able to provide informed written or verbal witnessed consent

Exclusion Criteria:

1. Patients receiving radical chemoradiation therapy (potentially curative and require parental feeding)
2. Have had more than one dose of new treatment.
3. Unstable acute condition (e.g., acute infection, severe uncontrolled symptoms) or
4. Underlying chronic condition (e.g., severe arthritis or dementia) that would impact study compliance.
5. Unable to provide written or verbal consent.
6. Insufficient English for consent and study procedures and appropriate interpretation unavailable

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | 24 weeks
  The Recruitment Rate will be assessed by the number of eligible patients approached vs the number of eligible patients consent for the study, providing a number of non-participations. This will be gathered as an aspect of feasibility.
Retention Rate | 24 weeks
  Retention rate will be examined via the number of those who consent to the study compared to the number of those who complete the study.
Secondary outcome data completion rate | 24 weeks
  Assessed by the total number of missing data from the total list of secondary outcomes
Rate of Intervention Completion | 12 weeks
  The percentage of exercises prescribed to the participants compared to the number of those completed.
Incidence of adverse effects and injuries related to the intervention | Week 1 to week 12
  Assessed by the number and rate of participant recorded adverse effects and injuries related to the intervention
Incidence of adverse events not related to the intervention | Week 1 to week 52
  The number of adverse events exhibited by the participants will be recorded with an associated grade (where relevant). A example list of adverse events are given below:
  * Constipation
  * Nausea
  * Vomiting
  * Diarrhoea
  * Skin Rash

SECONDARY OUTCOMES:
Free-living daily activity | Baseline, 24 weeks
  Accelerometer; the activpal4 micro units (activpal4; https://www.palt.com/pals/)
Australian Karnofsky Performance Scale (AKPS) | baseline, 12 and 24 weeks
  Single score from 10 to 100 (a higher score indicates better performance status).
Rockwood Frailty Index, a 7-point Clinical Frailty Scale | baseline, 12 and 24 weeks
  1 = very fit, and 7= severely frail.
Short Physical Performance Battery (SPBB) | baseline, 12 and 24 weeks
  Combines standing balance, 4 metre gait speed, and timed sit-to-stands to assess lower extremity function in older people
Grip strength | baseline, 12 and 24 weeks
  Maximum force/tension (kg) in the forearm muscles using a handheld dynamometer.
Bioelectrical impedance | baseline, 12 and 24 weeks
  Tanita body composition monitor and weight scale, a simple, non-invasive technique for measuring body composition in people with cancer
Weight (kg) | baseline, 12 and 24 weeks
  Tanita body composition monitor and weight scale
Patient-Generated Subjective Global Assessment (PG-SGA) | baseline and after 6, 12, and 24 weeks
  Assessment of nutritional status for people with cancer (scores from 0 - ≥9; 2-3 indicating need for basic nutrition intervention, 4-8 requiring dietetic intervention, and scores ≥9 indicating critical need for symptom management and nutritional intervention).
Community Healthy Activities Model Program for Seniors (CHAMPS) | baseline and after 6, 12, and 24 weeks
  Self-report total physical activity questionnaire designed to estimate weekly frequency of participation and energy expenditure in physical activities.
Integrated Patient Outcome Scale (IPOS) | baseline and after 6, 12, and 24 weeks
  measure of symptom burden with 20 items: one free-text question about main problems and concerns, 17 items on physical, psychological, spiritual problems, communication needs including with family, and practical support, scored on a 5-point Likert-type scale from 0 (best) to 4 (worst)
Client Service Receipt Inventory | baseline and after 6, 12, and 24 weeks
  Validated questionnaire designed to collect information on service utilisation, income, accommodation and other cost-related variables
EuroQol-5 Dimensions-5 Levels | baseline and after 6, 12, and 24 weeks
  The EQ-5D-5L is a generic health-related quality-of-life instrument with a descriptive system that comprises five dimensions (1) mobility, 2) self-care, 3) usual activities, 4) pain/discomfort, and 5) anxiety/depression), each of which has five levels of severity (given in statement form). Participants select a statement under each of the five dimensions which best suits their current state. In addition, the respiratory bolt on dimension for the EQ-5D-5L. For each dimension, lower scores indicate fewer problems in that domain (e.g. a score of 1 in mobility means no issues with mobility).
EuroQol-Visual Analogue Scale | baseline and after 6, 12, and 24 weeks
  The EQ-VAS is a self-report measure of overall health using a vertical visual analogue scale, ranging from 0 labelled as "worst possible" to 100 labelled as "best possible" health. Participants are then asked to write this number in a dedicated box.
Days alive and out of hospital | baseline, and after 6, 12, and 24 weeks
  Hospital admission (number of days) since starting the programme
Treatment completion rate | baseline, and after 6, 12, and 24 weeks
  Dose of cancer therapy received (percentage of dose received/dose prescribed) Treatment delay (days delayed)
Infection rate | baseline, and after 6, 12, and 24 weeks
  Assessed by the number of episodes requiring antibiotics (oral/IV) Number of episodes requiring hospital admission (number of days)
Treatment toxicity | baseline, and after 6, 12, and 24 weeks
  Cancer treatment-related toxicity (CTCAE v 5)
Height | baseline, 12 and 24 weeks
  measured in cm with a Seneca Stadiometer

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Forbes, PhD, Principal Investigator — Hull York Medical School, University of Hull
Locations (2):
- United Kingdom (2):
  - Hull University Teaching Hospitals NHS Trust, Hull, Yorkshire
  - York and Scarborough Teaching Hospitals NHS Trust, York, Yorkshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Swan F, Chen H, Forbes CC, Johnson MJ, Lind M. CANcer BEhavioural nutrition and exercise feasibility trial (CanBenefit); phase I qualitative interview findings. J Geriatr Oncol. 2021 May;12(4):641-648. doi: 10.1016/j.jgo.2020.09.026. Epub 2020 Oct 12. PMID 33059998
- [Result] Forbes CC, Swan F, Greenley SL, Lind M, Johnson MJ. Physical activity and nutrition interventions for older adults with cancer: a systematic review. J Cancer Surviv. 2020 Oct;14(5):689-711. doi: 10.1007/s11764-020-00883-x. Epub 2020 Apr 24. PMID 32328828